CLINICAL TRIAL: NCT06692660
Title: An Overview of the Use of Respiratory Support At Home in Children - Patients and Families Point of View
Brief Title: Overview: Use of Respiratory Support At Home in Children
Acronym: ELIPSE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A01045-42
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Sleep Apnea Syndromes in Children; Obesity in Children; Bronchopulmonary Dysplasia (BPD); Neuromuscular Disease; Storage Disease; Malformation; Alveolar Hypoventilation
Keywords: respiratory suport; sleep apnea syndrome; CPAP; BiPAP; ventilation; alveolar hypoventilation; non invasive ventilation
MeSH Terms: conditions — Pediatric Obesity; Bronchopulmonary Dysplasia; Neuromuscular Diseases; Congenital Abnormalities; Hypoventilation; Sleep Apnea Syndromes; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
the primary outcome is to describe the perceived success of the use of the respiratory support from the parent's point of view

DETAILED DESCRIPTION:
The use of ventilatory support, including CPAP (Continuous Positive Airway Pressure), which is a mode of ventilation with continuous positive pressure, and BiPAP (Bilevel Positive Airway Pressure), which is a mode of ventilation with two levels of pressure, has seen a significant increase in indications in recent years. The indications have become more numerous and increasingly complex. Sleep-related respiratory disorders, including obstructive sleep apnea-hypopnea syndrome, central apnea syndrome, and alveolar hypoventilation, are the primary reasons for these indications. In pediatrics, numerous conditions contribute to sleep-related respiratory disorders: ENT malformations, genetic conditions, obesity, bronchopulmonary dysplasia, neuromuscular diseases, thoracic deformities, and storage diseases.

The non-use or insufficient use of ventilatory support leads to a lack of treatment for sleep-related respiratory disorders. In the absence of treatment, the consequences are neurocognitive, cardiovascular, and metabolic, resulting in high morbidity. Non-use or insufficient use is a cause of failure of ventilatory support. Neither the use nor the failure of ventilatory support is clearly defined. It is crucial to evaluate the use of ventilatory support in order to correct factors related to non-use or insufficient use and to prevent the negative consequences resulting from unaddressed sleep-related respiratory disorders. This pilot study aims to assess the use of ventilatory support at home in pediatrics through interviews with patients and their parents. We will use a questionnaire designed for the study, consisting of 10 questions regarding sleep, symptoms, quality of life, technical issues, side effects, economic barriers, and adherence, to describe their experiences with ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* Children with respiratory support at home
* Age 0 to 18 (not yet passed) years old

Exclusion Criteria:

* Palliative care
* Invasive ventilation
* High flow oxygen therapy

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Our study population includes patients from the Grenoble Alpes Hospital, from 0 to 18 (not yet passed) years old. These patients benefit from respiratory support at home. Their follow-up is done at the Grenoble Alpes Hospital. We will not include patients who benefit from palliative care, invasive ventilation or high flow oxygen therapy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
describe the perceived success of the use of the respiratory support from the parent's point of view | Assessment during the filling of the questionnaire at enrollment
  The primary outcome measure is the median score and interquartile range, obtained from the answer modalities according to the Likert scale (scores ranging from 1 to 5), in response to the question from the parent interview guide, which states: "Do you consider that the ventilatory support proposed for your child is a success? Please circle the corresponding score."

SECONDARY OUTCOMES:
Describe the persistence of symptoms under ventilatory support according to the parent. | Assessment during the filling of the questionnaire at enrollment
  Answer to the question from the parent interview guide: "What symptoms did your child have before starting treatment? Have these symptoms improved?"
Describe the persistence of symptoms under ventilatory support according to the child | Assessment during the filling of the questionnaire at enrollment
  Answer to the question from the child interview guide: "Were you bothered before getting the machine? Is it better with the machine?"
Describe the tolerance of ventilatory support according to the parent. | Assessment during the filling of the questionnaire at enrollment
  Answer to the question from the parent interview guide: "Have you noticed any complications since your child started using the machine?"
Describe the tolerance of ventilatory support according to the child. | Assessment during the filling of the questionnaire at enrollment
  Answer to the question from the child interview guide: "Does the machine bother you?"
Describe adherence to ventilatory support according to the parent. | Assessment during the filling of the questionnaire at enrollment
  Answer to the question from the parent interview guide: "How many hours does your child use the machine at night? How many nights per week? Does your child use the machine when you go away for the weekend or on vacation...? If not, why?" For children aged 0-4 years: "Does the child wear it during naps? How many naps per week?"
Describe adherence to ventilatory support according to the child. | Assessment during the filling of the questionnaire at enrollment
  Answer to the question from the child interview guide: "Can you wear your machine all night? Every night? Do you wear your machine when you're not sleeping at home? If not, why? "

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble, Isère
  - Centre Hospitalier Grenoble Alpes, La Tronche

REFERENCES:
- [Background] Amaddeo A, Khirani S, Griffon L, Teng T, Lanzeray A, Fauroux B. Non-invasive Ventilation and CPAP Failure in Children and Indications for Invasive Ventilation. Front Pediatr. 2020 Oct 26;8:544921. doi: 10.3389/fped.2020.544921. eCollection 2020. PMID 33194886
- [Background] MacLean JE, Fauroux B. Long-term non-invasive ventilation in children: Transition from hospital to home. Paediatr Respir Rev. 2023 Sep;47:3-10. doi: 10.1016/j.prrv.2023.01.002. Epub 2023 Jan 12. PMID 36806331
- [Background] Ramirez A, Delord V, Khirani S, Leroux K, Cassier S, Kadlub N, Aubertin G, Picard A, Fauroux B. Interfaces for long-term noninvasive positive pressure ventilation in children. Intensive Care Med. 2012 Apr;38(4):655-62. doi: 10.1007/s00134-012-2516-1. Epub 2012 Mar 6. PMID 22392032
- [Background] McLaren AT, Bin-Hasan S, Narang I. Diagnosis, management and pathophysiology of central sleep apnea in children. Paediatr Respir Rev. 2019 Apr;30:49-57. doi: 10.1016/j.prrv.2018.07.005. Epub 2018 Jul 25. PMID 30170958
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Ramirez A, Khirani S, Aloui S, Delord V, Borel JC, Pepin JL, Fauroux B. Continuous positive airway pressure and noninvasive ventilation adherence in children. Sleep Med. 2013 Dec;14(12):1290-4. doi: 10.1016/j.sleep.2013.06.020. Epub 2013 Sep 25. PMID 24157098
- [Background] Bhattacharjee R, Benjafield AV, Armitstead J, Cistulli PA, Nunez CM, Pepin JD, Woehrle H, Yan Y, Malhotra A; medXcloud group. Adherence in children using positive airway pressure therapy: a big-data analysis. Lancet Digit Health. 2020 Feb;2(2):e94-e101. doi: 10.1016/S2589-7500(19)30214-6. Epub 2019 Dec 23. PMID 33334566
- [Background] Amaddeo A, Frapin A, Fauroux B. Long-term non-invasive ventilation in children. Lancet Respir Med. 2016 Dec;4(12):999-1008. doi: 10.1016/S2213-2600(16)30151-5. Epub 2016 Jul 13. PMID 27423917
- [Background] Fauroux B, Abel F, Amaddeo A, Bignamini E, Chan E, Corel L, Cutrera R, Ersu R, Installe S, Khirani S, Krivec U, Narayan O, MacLean J, Perez De Sa V, Pons-Odena M, Stehling F, Ferreira RT, Verhulst S. ERS statement on paediatric long-term noninvasive respiratory support. Eur Respir J. 2022 Jun 2;59(6):2101404. doi: 10.1183/13993003.01404-2021. Print 2022 Jun. PMID 34916265